CLINICAL TRIAL: NCT04260009
Title: An Open-Label, Phase 1/2 Dose Escalation and Expansion Trial to Evaluate the Pharmacokinetics, Safety, and Efficacy of Brigatinib as Monotherapy in Pediatric and Young Adult Patients With ALK+ Anaplastic Large Cell Lymphoma, Inflammatory Myofibroblastic Tumors or Other Solid Tumors
Brief Title: Pharmacokinetics, Safety, and Efficacy of Brigatinib Monotherapy in Pediatric and Young Adult Participants With ALK+ Anaplastic Large Cell Lymphoma, Inflammatory Myofibroblastic Tumors or Other Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reason unrelated to product safety
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Brigatinib-1002
Record Dates: First submitted 2020-01-22; First posted 2020-02-07 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Anaplastic Lymphoma Kinase Positive (ALK +) Anaplastic Large Cell Lymphoma; Inflammatory Myofibroblastic Tumors; Solid Tumors
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — brigatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Brigatinib (Experimental): Brigatinib tablet or age-appropriate formulation (AAF), orally once daily in 28-day Cycles with reference to adult dose of 90 mg in Week 1 and 180 mg starting in Week 2 based on participant's weight as dose level 1. Participants could receive dose level 2 based on safety and tolerability of dose level 1 in dose escalation phase (Ph).
  Interventions: Drug: Brigatinib; Drug: Brigatinib AAF
- Ph 2:Brigatinib (Unresectable/Recurrent ALK+ IMT) Participants (Experimental): Brigatinib recommended phase 2 dose (RP2D) determined during phase 1, tablet or AAF orally QD in participants with Unresectable/ Recurrent ALK+ IMT for up to 2 years in dose expansion phase.
  Interventions: Drug: Brigatinib; Drug: Brigatinib AAF
- Ph 2 :Brigatinib (Relapsed/Refractory ALK+ ALCL) Participants (Experimental): Brigatinib RP2D determined during phase 1, tablet or AAF orally QD in participants with Relapsed/ Refractory ALK+ ALCL for up to 2 years in dose expansion phase.
  Interventions: Drug: Brigatinib; Drug: Brigatinib AAF

INTERVENTIONS:
Drug: Brigatinib — Brigatinib tablets
Drug: Brigatinib AAF — Brigatinib age-appropriate formulation (AAF)

SUMMARY:
The purpose of this study is to estimate the maximum tolerated dose (MTD)/ recommended phase 2 dose (RP2D) regimen and characterize the pharmacokinetics (PK) of brigatinib monotherapy (film-coated tablets and age-appropriate formulation [AAF]) administered orally once daily (QD) in pediatric and young adult participants in Phase 1 and to define the efficacy of brigatinib administered as monotherapy within the disease-specific expansion arms (unresectable/recurrent anaplastic lymphoma kinase positive (ALK+) inflammatory myofibroblastic tumor (IMT); relapsed/refractory ALK+ anaplastic large cell lymphoma (ALCL) in Phase 2.

DETAILED DESCRIPTION:
The drug being tested in this study is called Brigatinib. Brigatinib is being tested to treat people who have Anaplastic Large Cell Lymphoma, Inflammatory Myofibroblastic Tumors or other solid tumours.

The study will enroll approximately 61 patients. Participants will be assigned to the following arm group to receive brigatinib:

* Phase 1 (Dose Escalation): Brigatinib Dose Level 1 and Dose Level 2 (based on safety and tolerability)
* Phase 2 (Dose Expansion): Unresectable/ Recurrent ALK+ IMT
* Phase 2 (Dose Expansion): Relapsed/ Refractory ALK+ ALCL

All participants will be administered brigatinib orally once daily in 28-day Cycles. Participants will receive fixed doses of brigatinib based on weight ranges. The starting doses in Phase 1 (Dose Level 1) are expected to provide systemic exposures of brigatinib in pediatric participants comparable to those achieved in adults receiving the recommended clinical dose of 90 mg once daily for 7 days followed by 180 mg once daily. One additional dose level (Dose Level 2) is planned in Phase 1 if the initial dose level is tolerated. This subsequent dose level is expected to provide systemic exposures of brigatinib in pediatric participants comparable to those achieved in adults receiving 90 mg once daily for 7 days followed by 240 mg once daily (the highest acceptably tolerated dose in adults). In Phase 2, brigatinib will be administered at the RP2D determined during Phase 1.

This multi-centre trial will be conducted worldwide. The overall time to participate in this study is approximately 36 months. Participants will make multiple visits to the clinic and will be contacted by telephone OR a final visit after receiving their last dose of brigatinib for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have confirmed cancer histologically or cytologically diagnosed at baseline
2. Participants are required to provide prior results showing an activating ALK aberration in the tumor (bone marrow aspirate, peripheral blood samples, biopsy, etc) documented by fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR) for the ALK-fusion transcript, next generation sequencing (NGS) or ALK immunohistochemistry (ALK immunohistochemistry can be used as a surrogate for FISH or NGS)
3. Phase 1, participants must be relapsed/refractory or intolerant to standard therapies or without option of established systemic therapy
4. Phase 2, participants must have measurable and/or evaluable disease:

   * Arm 1: IMT participants must not be suitable for curative surgical resection
   * Arm 2: participants must have relapsed/refractory ALCL
5. Performance Status: Karnofsky performance status ≥40% for participants >16 years of age or Lansky Play Scale ≥40% for participants ≤16 years of age
6. For participants receiving prior therapy:

   * Participants must have recovered to Grade <2 NCI CTCAE v5.0 or to baseline, from any nonhematologic toxicities (except alopecia and peripheral neuropathy) due to previous therapy
   * Participants who relapsed while receiving cytotoxic therapy: At least 14 days must have passed since the completion of the last dose of chemotherapy before the first dose of brigatinib can be given
   * Participants with hematologic malignancy and prior hematopoietic stem cell transplant (HSCT): Participants who have experienced relapse after a HSCT are eligible, provided they have no evidence of acute or chronic graft-versus-host disease (GVHD), are not receiving GVHD prophylaxis or treatment, and are at least 45 days posttransplant at the time of enrollment
   * Hematopoietic growth factors: Before the first dose of brigatinib, at least 7 days must have passed since completion of therapy with granulocyte colony-stimulating factor or other growth factors, and at least 14 days must have passed since completion of therapy with pegfilgrastim
   * Biologics and Targeted Therapies:

     * Immunotherapy: Before the first dose of brigatinib, at least 30 days must have passed after the completion of any type of immunotherapy, (eg, monoclonal antibodies [anti-PD1/PDL1], tumor vaccines, chimeric antigen receptor [CAR] T cells, etc.)
     * Other: before the first dose of brigatinib, at least 7 days must have passed since the last dose of a biologic agent. For agents that have known adverse events (AEs) occurring beyond 7 days after administration, this period must be extended beyond the time during which AEs are known to occur. The duration of this interval must be discussed with the sponsor's medical monitor/designee
   * Immunosuppressive therapy: Before the first dose of brigatinib, at least 14 days must have passed after the completion of immunosuppressive therapy (including regimens following stem cell transplant)
   * For symptomatic participants that urgently need relief (eg, airway obstruction), therapeutic doses of corticosteroids may be administered for a short course (up to 5 days)
   * Radiotherapy (XRT): No washout period is necessary for radiation given to any extramedullary site other than the CNS and lungs; ≥6 weeks must have passed if participants received prior total body irradiation or craniospinal or cranial XRT; ≥28 days must have passed if participants received radiotherapy to the lung(s)
7. Normal QT interval corrected per Fridericia method (QTcF) on screening electrocardiogram (ECG), defined as QTcF of ≤450 ms
8. Have life expectancy of ≥3 months.

Exclusion Criteria:

1. Participants receiving systemic treatment with strong or moderate cytochrome P450 3A (CYP3A) inhibitors or inducers within 14 days prior to the first dose of study drug
2. Previous treatment with brigatinib or other ALK inhibitors (except for participants in Phase 1)
3. Participants with completely resected stage-1 (ALCL and other lymphomas) disease
4. Participants with disease limited to skin (ALCL and other lymphomas)
5. Diagnosis of another concurrent primary malignancy
6. Clinically significant cardiovascular disease, including any of the following:

   * Myocardial infarction or unstable angina within 6 months of study entry
   * Uncontrolled hypertension defined as persistent elevation of systolic and/or diastolic blood pressures to ≥95th percentile based on age, sex, and height percentiles despite appropriate antihypertensive management
7. Planned non-protocol chemotherapy, radiation therapy, another investigational agent, or immunotherapy while participant is on study treatment
8. Uncontrolled seizure disorder. (Participants with seizure disorders that do not require antiepileptic drugs, or are well controlled with stable doses of antiepileptic drugs are eligible).
9. Any illness that affects gastrointestinal absorption
10. Ongoing or active systemic infection, active seropositive HIV, or known active hepatitis B or C infection.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) Regimen of Brigatinib Monotherapy | Up to 35 days
  MTD will be highest dose of brigatinib, at which <=1 of 6 participants would experience a dose-limiting toxicity (DLT). DLT is defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, as: Non-Haematological events possibly or definitively brigatinib related grade ≥3 AE except fatigue, nausea, vomiting lasting for <48 hours and nonhematologic laboratory abnormalities that resolve to Grade 1 or baseline within 7 days after study drug modification and/or supportive care; hematologic toxicities (except in participants with bone marrow involvement or MAS) as: Grade 4 neutropenia lasting longer than 7 days with supportive care, Grade ≥3 febrile neutropenia requiring antibiotics, Grade 3 platelet count (<50,000-25,000/μL) with bleeding requiring transfusion, Grade 4 platelet count (<25,000/μL) at any time, any delay or interruption of therapy of ≥2 weeks due to suspected treatment-related hematologic toxicities.
Phase 1: Recommended Phase 2 Dose (RP2D) of Brigatinib Monotherapy | Up to 35 days
  The RP2D is the maximum tolerated dose (MTD) or less. MTD was highest dose of Brigatinib, at which <=1 of 6 participants experienced DLT.
Phase 1: Maximum Observed Plasma Concentration (Cmax) of Brigatinib | Cycle 1, Days 1 and 15: Predose (Day 15 only) and at multiple timepoints (Up to 24 hours) post-dose; Predose on Day 1, Cycle 2 (each cycle is of 28 days)
Phase 1: Time of First Occurrence of Maximum Observed Plasma Concentration (Tmax) of Brigatinib | Cycle 1, Days 1 and 15: Predose (Day 15 only) and at multiple timepoints (Up to 24 hours) post-dose; Predose on Day 1, Cycle 2 (each cycle is of 28 days)
Phase 1: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Plasma Concentration (AUClast) of Brigatinib | Cycle 1, Days 1 and 15: Predose (Day 15 only) and at multiple timepoints (Up to 24 hours) post-dose; Predose on Day 1, Cycle 2 (each cycle is of 28 days)
Phase 2: Investigator-Confirmed Objective Response Rate (ORR) | Every 2 months until complete response is achieved (Up to 36 months)
  ORR is defined as the percentage of participants with tumor size reduction of a predefined amount and for a minimum time period. ORR is determined by radiological tests and investigator assessment. ORR for unresectable/recurrent ALK+IMT participants will be the achievement of a Complete Response (CR) or Partial Response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Per RECIST 1.1, CR is defined as disappearance of all target lesions; PR is defined as atleast 30% decrease in sum of diameters (SoD) of target lesions. Per International Pediatric Non-Hodgkin Lymphoma (IPNHL) response criteria, CR is defined as disappearance of all residual disease and tumor lesions; PR is defined as 50% decrease in sum of product of greatest perpendicular diameters (SPD) of lymphoma cells.

SECONDARY OUTCOMES:
Phase 1: Number of Participants with Dose Limiting Toxicity (DLTs) | Up to 35 days
  DLT is defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, as: Non-Haematological events possibly or definitively brigatinib related grade ≥3 AE except fatigue, nausea, vomiting lasting for <48 hours and nonhematologic laboratory abnormalities that resolve to Grade 1 or baseline within 7 days after study drug modification and/or supportive care; hematologic toxicities (except in participants with bone marrow involvement or MAS) as: Grade 4 neutropenia lasting longer than 7 days with supportive care, Grade ≥3 febrile neutropenia requiring antibiotics, Grade 3 platelet count (<50,000-25,000/μL) with bleeding requiring transfusion, Grade 4 platelet count (<25,000/μL) at any time, any delay or interruption of therapy of ≥2 weeks due to suspected treatment-related hematologic toxicities.
Phases 1 and 2: Percentage of Participants With One or More Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose of study drug up to 30 days after last dose of study drug (Up to approximately 2 years)
  An AE is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. A SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Overall Acceptability and Palatability as Assessed by Acceptability and Palatability Questionnaire Score | Days 1 and 8 (Cycle 1)
  Acceptability is defined as the overall ability of the participant to use the medicine as intended. Acceptability and palatability (taste and smell) will be assessed using a 5-point facial hedonic scale, where 1 indicates 'bad', and 5 indicates 'good'.
Phase 2: Duration of Response (DOR) | From the first dose of study drug up to disease progression or death (Up to 36 months)
  DOR is defined as the time from the initial assessment of CR response until subsequent disease progression or relapse. Per RECIST 1.1, CR is defined as disappearance of all target lesions and per IPNHL, response criteria CR is defined as disappearance of all residual disease and tumor lesions. Disease progression as per RECIST 1.1, is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Disease progression as per IPNHL response criteria, is defined as development of new morphologic evidence of disease in bone marrow.
Phase 2: Time to Response | From the first dose of study drug up to disease progression or death (Up to 36 months)
  Time from the start of treatment with brigatinib to the first objective tumor response observed for participants who achieved a CR or PR. Per RECIST 1.1, CR is defined as disappearance of all target lesions; PR is defined as atleast 30% decrease in sum of diameters (SoD) of target lesions. Per IPNHL response criteria, CR is defined as disappearance of all residual disease and tumor lesions; PR is defined as 50% decrease in sum of product of greatest perpendicular diameters (SPD) of lymphoma cells.
Phase 2: Disease Control Rate in Unresectable/ Recurrent ALK+ IMT Participants | From the first dose of study drug up to disease progression or death (Up to 36 months)
  DCR is defined as the percentage of participants who are confirmed to have achieved CR or PR or have a best overall response of stable disease (SD). Per RECIST 1.1, CR is defined as disappearance of all target lesions; PR is defined as atleast 30% decrease in sum of diameters (SoD) of target lesions. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Phase 2: Progression Free Survival (PFS) in Unresectable/ Recurrent ALK+ IMT Participants | From the first dose of study drug up to disease progression or death (Up to 36 months)
  PFS is defined as the time from the date of first dose to the date of PD per RECIST v1.1, or the date of death due to any cause, whichever occurs first. PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Phase 2: Event-free Survival in Relapsed/ Refractory ALK+ ALCL Participants | From the first dose of study drug up to disease progression or death (Up to 36 months)
  EFS is defined as the time from the date of first dose to any treatment failure including disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death). Participants without any treatment failure events will be censored at last known alive date before data cutoff date.
Phase 2: Overall Survival | Up to 36 months
  Overall survival in months is defined as the time from the date of first dose to the date of death due to any cause. Participants without documentation of death at the time of analysis will be censored at the date last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.